CLINICAL TRIAL: NCT05725460
Title: Efficacy of Dextrose 5% in Comparison With Steroid in Median Nerve Ultrasound Guided Hydrodissection in Patients With Carpal Tunnel Syndrome
Brief Title: Ultrasound Guided Median Nerve Hydrodissection Using Dextrose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iraqi Board of medical specialties (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iraqiboard
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-05

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: 2 groups comparing the efficacy of dextrose water 5 % in median nerve hydrodissection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dextrose 5% (Experimental): 10 mls of dextrose under ultrasound to separate the median nerve from adjacent structures
  Interventions: Procedure: dextrose 5% median nerve hydrodissection
- steroid (Active Comparator): 10 mls of steroid used to separate the median nerve from adjacent structures
  Interventions: Procedure: dextrose 5% median nerve hydrodissection

INTERVENTIONS:
Procedure: dextrose 5% median nerve hydrodissection — planned to be a good alternative to steroid hydrodissection

SUMMARY:
to compare the efficacy of dextrose 5% with steroid hydrodissection in patients with carpal tunnel syndrome

DETAILED DESCRIPTION:
in some cases there is prohibition to use steroid with example the patient rejection to use steroid the maneuver planned median nerve hydrodissection using ultrasound and 10 mld of dextrose 5%, unleash the median nerve for the surrounding structure and short follow up planned to be 2 weeks

ELIGIBILITY:
Inclusion Criteria:

severe carpal tunnel syndrome failed medical management -

Exclusion Criteria:

previous failed surgery previous failed injection previous failed trial of hydrodissection cervical or brachial nerve entrapment wrist osteoarthritis or rheumatoid pregnant diabetes mellitus

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
pain relief in 2 weeks follow up | 6 months
  difference in sensory and functional symptoms post median nerve hydrodissection using dextrose and compare this effect with steroid population arm using Boston questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad Medical City, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided